CLINICAL TRIAL: NCT04278664
Title: Effect of Telemedicine on Outcomes in Pregnant Women With Type 1 Diabetes Mellitus
Brief Title: Telemedicine in Pregnant Women With Type 1 Diabetes Mellitus
Status: Terminated | Type: Observational
Why Stopped: low enrollment
Sponsor: Ana Braescu (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor-Investigator, Ana Braescu, Research Coordinator, Pediatrix
Organization: Pediatrix (Other)
Other Study IDs: 1506903391 UA IRB#
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes; Pregnancy in Diabetic
Keywords: telemedicine; Type 1 diabetes in pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesize that co-managing pregnant type 1 diabetics with telemedicine will have at least equivalent outcomes to those managed with standard care. Comparison of outcomes between pregnant type 1 diabetics being co-managed with telemedicine compared to those receiving conventional care will help identify unanswered clinical questions and areas for improvement in regard to standards of care for pregnant type 1 diabetics. The data generated from this analysis will help determine whether telemedicine can be an effective additional means of care for pregnant type 1 diabetic patients.

DETAILED DESCRIPTION:
Few studies have researched the use of telemedicine in the management of type 1 diabetes during pregnancy. These studies are additionally limited due to the number of patients as well as several secondary outcomes reported. Therefore, this study will enroll 100 participants to reach a power of 81.8% with HbA1c as a primary outcome and secondary outcomes related to diabetic management such as frequency of hypoglycemia, antenatal hospital stay (percentage requiring admission, length of stay), miscarriage, cesarean section rates, induction of labor, fetal birth weight, gestational age at birth or preterm birth (<34 weeks, <37 weeks), frequency of neonatal hypoglycemia, shoulder dystocia, neonatal death, major and minor anomalies, and neonatal intensive care admission.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetics who are at or less than 16 weeks in their pregnancy
* 18 years of age or more
* Voluntary participation

Exclusion Criteria:

* <18 years of age
* Not Type I diabetic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Maternal glycemic control in Type I Diabetics during pregnancy will be studied by enrolling patients in two different groups: one will be treated with the current standard of care for a type 1 diabetic pregnancy and the other group will receive the same standard of care in addition to utilizing telemedicine communication of glucose and insulin readings during weeks when there are no recommended physician visits. All participants will be monitored throughout their pregnancy and clinical outcomes will be reviewed upon delivery and a 6-week postpartum visit. This study is important in adding to current literature regarding the role of telemedicine in pregnant type 1 diabetic care as it could potentially lead to changes in the current standard care for pregnant type 1 diabetics.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
HbA1c, maternal glycemic control | first trimester in pregnancy through 6 weeks postpartum
  maternal glycemic control during pregnancy as measured by HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: C. Kevin Huls, MD, Principal Investigator — Pediatrix

IPD SHARING:
Plan to Share IPD: No